CLINICAL TRIAL: NCT06534437
Title: An Open Label, Phase 2 Clinical Trial of MEN1703 as Monotherapy and in Combination With Glofitamab in Patients With Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphoma
Brief Title: MEN1703 (SEL24) to Treat Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphoma (JASPIS-01)
Acronym: JASPIS-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryvu Therapeutics SA (Industry)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JASPIS-01
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Non-Hodgkin Lymphoma, B-cell
Keywords: Relapsed; Refractory; Aggressive
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence; Aggression | interventions — glofitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MEN1703 + glofitamab (Experimental): • Participants who are naïve to treatment with an anti-CD3xCD20 bispecific antibody (group 1) will be given MEN1703 orally at a dose of 150 mg daily for 7 days or 125 mg daily for 14 days, in 21-day cycles for a maximum of 12 cycles, in combination with glofitamab administered as an IV infusion in a step-up dosing schedule starting with 2.5 mg on day 8 of cycle 1, and10 mg on day 15 of cycle 1, and 30 mg on day 1 from cycle 2 onward until disease progression or withdrawal, for a maximum of 12 cycles (parts 1, 2, 3)).
  All participants will be administered 1,000 mg of obinutuzumab as an IV infusion on cycle 1 day 1.
  • Participants who have exhausted all standard treatment options (group 2) will receive MEN1703 as a single-agent, at a dose of 125 mg orally every-day for 14 consecutive days in consecutive 21-day treatment cycles, until progressive disease (parts 1 and 2).
  Interventions: Drug: MEN1703; Drug: Glofitamab
- Gofitamab (Active Comparator): Participants who are naïve to treatment with an anti-CD3xCD20 bispecific antibody (group 1) will receive glofitamab as a single-agent administered as an IV infusion in a step-up dosing schedule starting with 2.5 mg on day 8 of cycle 1, and10 mg on day 15 of cycle 1, and 30 mg on day 1 from cycle 2 onward until disease progression or withdrawal, for a maximum of 12 cycles (part 3).
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: MEN1703 — MEN1703 (Dapolsertib hydrochloride) is a potent dual inhibitor of proviral integration site for Moloney murine leukemia virus (PIM) kinases and Fms-like tyrosine kinase 3 (FLT3).
  Other Names: SEL24; Dapolsertib hydrochloride
  Arms: MEN1703 + glofitamab
Drug: Glofitamab — Glofitamab is a bispecific monoclonal antibody that binds bivalently to CD20 expressed on the surface of B-cells and monovalently to CD3 in the T-cell receptor complex expressed on the surface of T-cells.

SUMMARY:
The goal of the study is to assess the safety and anti-lymphoma activity of MEN1703 (Dapolsertib hydrochloride) when given as a single-agent or combined with glofitamab to patients with relapsed/refractory (R/R) aggressive B-cell non-Hodgkin lymphoma. The study will be open to groups at the same time:

* Group 1 - patients who have not had anti-CD3xCD20 bispecific antibody therapy but who have had at least 2 prior lines of systemic treatment for aggressive B-cell non-Hodgkin lymphoma
* Group 2 - patients who have exhausted all standard treatment options including at least 2 prior lines of systemic treatment for aggressive B-cell non-Hodgkin lymphoma Group 1 patients will be treated for a maximum of 12 cycles. One cycle is 21 days. Group 2 with be treated until the disease progresses, therefore treatment duration is dependent on the number of treatment cycles a participant receives prior to progression.

DETAILED DESCRIPTION:
The study consists of 3 parts, to investigate MEN1703 (Dapolsertib hydrochloride) in combination with glofitamab in patients who are naïve to treatment with an anti-CD3xCD20 bispecific antibody (group 1) or MEN1703 alone in patients who have exhausted all standard treatment options (group 2).

Part 1 (safety run-in) and Part 2 (enrichment): patients who are naïve to treatment with an anti-CD3xCD20 bispecific antibody (group 1) will receive either 150 mg or 125 mg of MEN1703 along with glofitamab. Patients who have exhausted all standard treatment options (group 2) will receive 125 mg of MEN1703 as a single-agent.

Part 3 (optional randomized comparison): Patients who are naïve to treatment with an anti-CD3xCD20 bispecific antibody therapy will be randomized to receive either MEN1703 (Dapolsertib hydrochloride) at a dose selected from part 2 in combination with glofitamab or glofitamab alone.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Documented histological confirmation of aggressive B-cell non-Hodgkin lymphoma including DLBCL NOS and transformed indolent B-cell lymphoma
3. Relapsed or refractory disease having received at least 2 prior lines of systemic treatment and, naïve to anti-CD3xCD20 bispecific antibody treatment (group 1) or exhausted all standard, available treatment options (group 2)
4. At least 1 measurable site of disease based on computed tomography (CT) or positron emission tomography (PET)-CT scan with involvement of 2 or more clearly demarcated lesions and or nodes.
5. Availability of lymph node tissue at Screening (or archival sample) (part 2 participants only)
6. Life expectancy of ≥12 weeks.
7. Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
8. Adequate organ function at Screening
9. Adequate hematologic function

Exclusion Criteria:

1. Primary central nervous system (CNS) lymphoma or CNS involvement by lymphoma at screening.
2. Received anti-cancer treatments, including cytotoxic chemotherapy, radiotherapy, hormonal therapy, biologic, immunotherapy, or investigational drugs within 14 days or 5 half-lives (whichever is shorter) before the first dose of study drug. Prior treatment with CAR-T cell or an anti-CD3xCD20 bispecific antibody therapy (permitted for Group 2 only), requires a wash out period of ≥4 weeks.
3. Concurrent participation in another therapeutic clinical study.
4. Ongoing clinically significant toxicity (for example, alopecia is not clinically significant) from any prior anti-cancer therapy that has not resolved to Grade 1 or less prior to the first dose of study drug.
5. Prior treatment with a PIM inhibitor.
6. Group 1 only: Any prior therapy with a bispecific antibody targeting CD3 and CD20.
7. Known risk of allergy to the study drugs, MEN1703 (group 1 and 2) or glofitamab (group 1) or their excipients
8. Contraindication to all uric acid lowering agents.
9. Major surgery within 1 month prior to first dose of study drug.
10. Hematopoietic stem cell transplant within 4 months prior to first dose of study drug.
11. Requires systemic immune-modulating therapy (regardless of dose) or has confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression.
12. Exposed to live or live attenuated vaccine(s) within 4 weeks prior to signing the informed consent form (ICF).
13. Evidence of ongoing and uncontrolled systemic bacterial, fungal, or viral infection, except for documented Grade Common Terminology Criteria for Adverse Events (CTCAE) ≤2 infections with evidence of improvement or without evidence of worsening infection.
14. Known human immunodeficiency virus (HIV) infection
15. Current active liver disease from any cause
16. Ongoing drug-induced pneumonitis.
17. Ongoing inflammatory bowel disease.
18. Active known second malignancy
19. Received an agent known to be a sensitive CYP2D6 substrate or a CYP2D6 substrate with a narrow therapeutic range, a strong or moderate CYP2D6 inhibitor, or a BCRP inhibitor within 14 days or 5 half-lives (whichever is shorter), prior to the first dose of study drug.
20. Cardiac dysfunction is defined as myocardial infarction within 6 months of study entry, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled dysrhythmias, or poorly controlled angina.
21. Receiving treatment for active, ongoing thromboembolic event. Note: Does not apply to prophylactic treatment to prevent or avoid reoccurrence of a prior resolved event. To review with Medical Monitor where further risk assessment is needed.
22. History of serious ventricular arrhythmia (e.g., VT or VF, ≥3 beats in a row), or QT interval corrected for heart rate (QTc) ≥480 ms.

    Note: QTc values up to 500 ms will be acceptable where patient's medical history e.g., bundle branch block, is known to cause mild QTc prolongation and the condition is well controlled.
23. Any disease, syndrome or condition which may significantly affect drug intake via oral route.
24. Planning to become pregnant or breastfeed during treatment and for 1 month after the last dose of study drug.
25. Any other prior or current medical condition, intercurrent illness, surgical history, physical or 12-lead electrocardiogram (ECG) findings, laboratory abnormalities, or extenuating circumstance (e.g., alcohol or drug addiction) that, in the investigator's opinion, could jeopardize patient safety or interfere with the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence and severity of adverse events (AE) | 12 months
  Assessed as the number and grade of adverse events assessed by CTCAE v5.0
Part 2 and Part 3: Complete response (CR) (group 1) | 12 months
  Assessed per Lugano Response Criteria for Malignant Lymphoma
Part 2 and Part 3: Overall response rate (group 2) | 12 months
  Assessed as the number of patients who achieve a complete response (CR) or partial response (PR), per Lugano Response Criteria, divided by the total number of evaluable patients

SECONDARY OUTCOMES:
Part 2 and Part 3, Incidence and severity of AE | 12 months
  Assessed as the number and grade of adverse events assessed by CTCAE v5.0
Maximum Plasma Concentration (Cmax) | 12 months
  Assessment of the peak plasma concentration (Cmax)
Maximum Plasma Concentration (Tmax) | 12 months
  Assessment of the time to peak plasma concentration (Tmax)
Area Under the Concentration Time-Curve (AUC) | 12 months
  Assessed of the area under the plasma concentration versus time curve (AUC)
Impact of treatment on patient reported outcomes (PRO) | 12 months
  Assessed as changes in lymphoma symptoms, well-being, and general health status measured according to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) consisting of 30 questions that assess five domains of patient functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), global health status/quality of life (GHS/QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All are scored from 0 to 100, with higher scores on the five domains and GHS/QoL being reflective of better health related (HR) QoL, and higher scores on the symptom scales and single items reflective of poor HRQoL.
Impact of treatment on quality of life (QOL) | 12 months
  Assessed as changes in lymphoma symptoms and health related quality of life (HRQoL) as measured using the 15-item Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) including physical, social/family, emotional, and functional well-being and includes a lymphoma-specific subscale. The scale range is 0 to 60, with a higher score reflecting a better HRQoL.
Overall survival (OS) | 12 months
  Assessed as the time from first treatment to death.
Progression-free survival (PFS) | 12 months
  Assessed as time from the time from first treatment to the first occurrence of disease progression or death.
Duration of Response (DoR) | 12 months
  Assessed as the time from first response (CR or PR) to the first occurrence of disease progression or death.
Duration of Complete Response (DoCR) | 12 months
  Assessed as the time from first complete response (CR) to the first occurrence of disease progression or death.
Time to response | 12 months
  Assessed as the time from the first treatment to the time of first response (CR or PR).
Time to next treatment | 12 months
  Assessed as the time from the first treatment to the start date of the first therapy received after the participant has ended study treatment and received subsequent anti-lymphoma therapy.

CONTACTS AND LOCATIONS:
Locations (36):
- France (7):
  - Centre Hospitalier Le Mans, Le Mans
  - CHU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Limoges - CHU Dupuytren, Limoges
  - Hospices Civils De Lyon - Hôpital Lyon Sud, Lyon
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - APHP - Hôpital Pitié-Salpêtrière, Paris
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
- Poland (13):
  - Wojewódzki Szpital Specjalistyczny w Białej Podlaskiej, Biała Podlaska
  - IN-VIVO Bydgoszcz Sp. z o.o., Bydgoszcz
  - Klinika Hematologii I Transplantologii Uck, Gdansk
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej Curie, Państwowy Instytut Badawczy, Gliwice
  - Pratia Hematologia Sp. z o.o., Katowice
  - Pratia MCM Kraków, Krakow
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Aidport Sp. z o.o., Skórzewo
  - Wojewódzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Lux Med Onkologia Sp. z o.o., Warsaw
  - Wojskowy Instytut Medyczny - Państwowy Instytut Badawczy, Warsaw
- Spain (10):
  - Hospital Universitari Vall D Hebron, Barcelona
  - Clinica Universidad De Navarra, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Hospital Clínico Uni versitario Virgen de la Arrixaca, Murcia
  - Clinica Universidad De Navarra, Pamplona
  - Hospital Universitario De Navarra, Pamplona
  - Hospital Universitario De Salamanca, Salamanca
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- United Kingdom (6):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Royal Marsden Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Plymouth Hospitals NHS Trust, Plymouth
  - The Royal Marsden Hospital, Sutton
  - St George's Hospital, Tooting

IPD SHARING:
Plan to Share IPD: No